CLINICAL TRIAL: NCT03866837
Title: Prebiotic GOS and Lactoferrin for Beneficial Gut Microbiota With Iron Supplements
Brief Title: Prebiotic GOS and Lactoferrin With Iron Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Swiss Federal Institute of Technology (Other); Jomo Kenyatta University of Agriculture and Technology (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Gary M Brittenham, MD, Professor of Pediatrics and Medicine, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAR8900; R01DK115449 (NIH)
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Iron-deficiency
Keywords: Iron-deficiency; Iron supplementation; Galacto-oligosaccharides; Lactoferrin; Ferrous fumarate; Clinical trial; Microbiome; PolyFermS; Polyfermenter intestinal model
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron

STUDY DESIGN:
Intervention Model Description: The study is a single-center, double-blinded, randomized, 9-month clinical trial with a 2X2 factorial design to determine the efficacy of galacto-oligosaccharides and bovine lactoferrin in preserving a beneficial gut microbiota during iron supplementation in Kenyan infants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stratified randomization will be carried out by the Trial Statistician using computer-generated randomly permuted blocks of size 2, 4 or 6 with stratification by gender and assignment of eligible infants to one of the 4 intervention groups using 4 color codes. Allocation will be known solely by the Trial Statistician and the Clinical Trial Safety Officer and concealed from all other study personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study group A: GOS (Active Comparator): This study group will receive daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]) and galacto-oligosaccharides (GOS), 7.5 mg.
  Interventions: Dietary Supplement: Galacto-oligosaccharides; Dietary Supplement: Multiple micronutrient powders with 5 mg iron
- Study group B: bLF (Active Comparator): This study group will receive daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]), bovine lactoferrin (bLF), 1.0 g.
  Interventions: Dietary Supplement: Bovine lactoferrin; Dietary Supplement: Multiple micronutrient powders with 5 mg iron
- Study group C: GOS + bLF (Active Comparator): This study group will receive daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]), galacto-oligosaccharides (GOS), 7.5 mg, and bovine lactoferrin (bLF), 1.0 g.
  Interventions: Dietary Supplement: Galacto-oligosaccharides; Dietary Supplement: Bovine lactoferrin; Dietary Supplement: Multiple micronutrient powders with 5 mg iron
- Study group D (Placebo Comparator): This study group will receive daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]) alone, with no galacto-oligosaccharides (GOS), and no bovine lactoferrin (bLF).
  Interventions: Dietary Supplement: Multiple micronutrient powders with 5 mg iron

INTERVENTIONS:
Dietary Supplement: Galacto-oligosaccharides — Galacto-oligosaccharides are classified as Generally Recognized As Safe (GRAS) by the U.S. Food and Drug Administration, are components of cow's milk and have been used repeatedly in clinical trials without adverse effects.
  Arms: Study group A: GOS; Study group C: GOS + bLF
Dietary Supplement: Bovine lactoferrin — Bovine lactoferrin is classified as Generally Recognized As Safe (GRAS) by the U.S. Food and Drug Administration, is a component of cow's milk and has been used repeatedly in clinical trials without adverse effects.
  Arms: Study group B: bLF; Study group C: GOS + bLF
Dietary Supplement: Multiple micronutrient powders with 5 mg iron — The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].

SUMMARY:
The ultimate goal of this research is to develop a means to safely administer iron supplements to infants in settings with a high infection burden. The investigators will conduct a randomized clinical trial in 6 month-old Kenyan infants in conjunction with mechanistic microbiota studies using a novel long-term continuous polyfermenter platform inoculated with immobilized fecal microbiota from Kenyan infants. Oral iron supplements are associated with a significant 15% increase in the rate of diarrhea in children in malaria-endemic areas. The most recent studies have shown that prebiotic galacto-oligosaccharides (GOS) can provide partial amelioration of the adverse effects of iron supplementation by enhancing the growth of barrier populations of bifidobacteria and lactobacilli. The investigators hypothesize that the combination of GOS with bovine lactoferrin, adding iron sequestration as well as antimicrobial and immunomodulatory activities, will provide almost complete protection against the adverse effects of added iron on the intestinal microbiota.

DETAILED DESCRIPTION:
Iron deficiency, the principal cause of anemia globally, affects more than two billion individuals, predominantly infants, children and women of childbearing age. Iron deficiency impairs cognitive and behavioral development in childhood, compromises immune responsiveness, decreases physical performance, and when severe, increases mortality among infants, children and pregnant women. Effective prevention and treatment of iron deficiency uses iron supplements or fortificants to increase oral iron intake. Generally, only a small fraction of the added iron is absorbed in the upper small intestine, with 80% or more passing into the colon. Because iron is an essential micronutrient for growth, proliferation, and persistence for most intestinal microbes, the increase in iron availability has profound effects on the composition and metabolism of intestinal microbiota. In particular, iron is a prime determinant of colonization and virulence for most enteric gram-negative bacteria, includingmSalmonella, Shigella and pathogenic Escherichia coli. Commensal intestinal microorganisms, principally of the genera Bifidobacterium and Lactobacillus, require little or no iron, provide a barrier effect and can inhibit pathogen growth by a variety of methods, including sequestration of iron, competition for nutrients and for intestinal epithelial sites stabilization of intestinal barrier function, and production of antibacterial peptides and organic acids that lower the pH. Increases in unabsorbed iron can promote the growth of virulent enteropathogens that overwhelm barrier strains and disrupt the gut microbiota.

We hypothesize that the combination of prebiotic GOS with bovine lactoferrin (bLF), adding iron sequestration, antimicrobial and immunomodulatory activities, will provide virtually complete protection against the adverse effects of added iron on the intestinal microbiota. Our research has two specific aims:

1. to conduct a randomized, controlled double-blind 9-month clinical trial in 6-month old Kenyan infants comparing the effects on gut microbiome composition among groups receiving in-home fortification for 6 months with micronutrient powders containing 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]) and (i) galacto-oligosaccharides (GOS; 7.5 g), (ii) bovine lactoferrin (bLF, 1.0 g), (iii) GOS (7.5 g) and bLF (1.0 g), and (iv) no GOS or bLF. Each infant will then be followed for an additional 3 months to determine the longer-term effects of the treatments.
2. to examine mechanisms of iron, prebiotic GOS and iron-sequestering bLF on microbiota composition, enteropathogen development, microbiota functions and metabolic activity, and inflammatory potential in vitro with treatments paralleling those in Specific Aim 1, using immobilized fecal microbiota from Kenyan infants to inoculate our established long-term continuous polyfermenter intestinal model (PolyFermS) to mimic Kenyan infant colon conditions, together with cellular studies.

Combining in vivo clinical and in vitro approaches will help guide formulation of safer iron supplements and fortificants and improve our understanding of the mechanisms whereby prebiotic GOS and iron-sequestering bLF support commensal microbiota to prevent iron-induced overgrowth by opportunistic enteropathogens.

ELIGIBILITY:
Inclusion Criteria:

* vaginal or cesarean delivery
* an infant age of 6 months (±3 weeks)
* mother ≥15 years of age
* infant still breastfeeding
* anticipated residence in the area for the study duration.

Exclusion Criteria:

* inability to provide informed consent
* hemoglobin < 70 g/L
* Z scores for weight-for-age (WAZ) or weight-for-height (WHZ) <3,
* any maternal or infant chronic illness
* administration of any infant vitamin or mineral supplements for the past 2 months
* history of infant antibiotic treatment within 7 days before study enrollment.

Ages: 21 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Brittenham, MD, Principal Investigator — Columbia University
Locations (2):
- Jomo Kenyatta University of Agriculture and Technology, Nairobi, Kenya
- Swiss Federal Institute of Technology (ETH Zürich), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaeggi T, Kortman GA, Moretti D, Chassard C, Holding P, Dostal A, Boekhorst J, Timmerman HM, Swinkels DW, Tjalsma H, Njenga J, Mwangi A, Kvalsvig J, Lacroix C, Zimmermann MB. Iron fortification adversely affects the gut microbiome, increases pathogen abundance and induces intestinal inflammation in Kenyan infants. Gut. 2015 May;64(5):731-42. doi: 10.1136/gutjnl-2014-307720. Epub 2014 Aug 20. PMID 25143342
- [Background] Paganini D, Uyoga MA, Zimmermann MB. Iron Fortification of Foods for Infants and Children in Low-Income Countries: Effects on the Gut Microbiome, Gut Inflammation, and Diarrhea. Nutrients. 2016 Aug 12;8(8):494. doi: 10.3390/nu8080494. PMID 27529276
- [Background] Zimmermann MB, Chassard C, Rohner F, N'goran EK, Nindjin C, Dostal A, Utzinger J, Ghattas H, Lacroix C, Hurrell RF. The effects of iron fortification on the gut microbiota in African children: a randomized controlled trial in Cote d'Ivoire. Am J Clin Nutr. 2010 Dec;92(6):1406-15. doi: 10.3945/ajcn.110.004564. Epub 2010 Oct 20. PMID 20962160
- [Background] Dostal A, Chassard C, Hilty FM, Zimmermann MB, Jaeggi T, Rossi S, Lacroix C. Iron depletion and repletion with ferrous sulfate or electrolytic iron modifies the composition and metabolic activity of the gut microbiota in rats. J Nutr. 2012 Feb;142(2):271-7. doi: 10.3945/jn.111.148643. Epub 2011 Dec 21. PMID 22190022
- [Background] Dostal A, Fehlbaum S, Chassard C, Zimmermann MB, Lacroix C. Low iron availability in continuous in vitro colonic fermentations induces strong dysbiosis of the child gut microbial consortium and a decrease in main metabolites. FEMS Microbiol Ecol. 2013 Jan;83(1):161-75. doi: 10.1111/j.1574-6941.2012.01461.x. Epub 2012 Aug 28. PMID 22845175
- [Background] Dostal A, Lacroix C, Pham VT, Zimmermann MB, Del'homme C, Bernalier-Donadille A, Chassard C. Iron supplementation promotes gut microbiota metabolic activity but not colitis markers in human gut microbiota-associated rats. Br J Nutr. 2014 Jun 28;111(12):2135-45. doi: 10.1017/S000711451400021X. Epub 2014 Feb 21. PMID 24555487
- [Background] Dostal A, Gagnon M, Chassard C, Zimmermann MB, O'Mahony L, Lacroix C. Salmonella adhesion, invasion and cellular immune responses are differentially affected by iron concentrations in a combined in vitro gut fermentation-cell model. PLoS One. 2014 Mar 27;9(3):e93549. doi: 10.1371/journal.pone.0093549. eCollection 2014. PMID 24676135
- [Background] Dostal A, Lacroix C, Bircher L, Pham VT, Follador R, Zimmermann MB, Chassard C. Iron Modulates Butyrate Production by a Child Gut Microbiota In Vitro. mBio. 2015 Nov 17;6(6):e01453-15. doi: 10.1128/mBio.01453-15. PMID 26578675
- [Background] Lacroix C, de Wouters T, Chassard C. Integrated multi-scale strategies to investigate nutritional compounds and their effect on the gut microbiota. Curr Opin Biotechnol. 2015 Apr;32:149-155. doi: 10.1016/j.copbio.2014.12.009. Epub 2015 Jan 3. PMID 25562815
- [Background] Payne AN, Zihler A, Chassard C, Lacroix C. Advances and perspectives in in vitro human gut fermentation modeling. Trends Biotechnol. 2012 Jan;30(1):17-25. doi: 10.1016/j.tibtech.2011.06.011. Epub 2011 Jul 20. PMID 21764163
- [Background] Payne AN, Chassard C, Banz Y, Lacroix C. The composition and metabolic activity of child gut microbiota demonstrate differential adaptation to varied nutrient loads in an in vitro model of colonic fermentation. FEMS Microbiol Ecol. 2012 Jun;80(3):608-23. doi: 10.1111/j.1574-6941.2012.01330.x. Epub 2012 Mar 27. PMID 22324938
- [Background] Tanner SA, Zihler Berner A, Rigozzi E, Grattepanche F, Chassard C, Lacroix C. In vitro continuous fermentation model (PolyFermS) of the swine proximal colon for simultaneous testing on the same gut microbiota. PLoS One. 2014 Apr 7;9(4):e94123. doi: 10.1371/journal.pone.0094123. eCollection 2014. PMID 24709947
- [Background] Zihler Berner A, Fuentes S, Dostal A, Payne AN, Vazquez Gutierrez P, Chassard C, Grattepanche F, de Vos WM, Lacroix C. Novel Polyfermentor intestinal model (PolyFermS) for controlled ecological studies: validation and effect of pH. PLoS One. 2013 Oct 30;8(10):e77772. doi: 10.1371/journal.pone.0077772. eCollection 2013. PMID 24204958
- [Background] Pasricha SR, Hayes E, Kalumba K, Biggs BA. Effect of daily iron supplementation on health in children aged 4-23 months: a systematic review and meta-analysis of randomised controlled trials. Lancet Glob Health. 2013 Aug;1(2):e77-e86. doi: 10.1016/S2214-109X(13)70046-9. Epub 2013 Jul 24. PMID 25104162
- [Background] Kassebaum NJ, Jasrasaria R, Naghavi M, Wulf SK, Johns N, Lozano R, Regan M, Weatherall D, Chou DP, Eisele TP, Flaxman SR, Pullan RL, Brooker SJ, Murray CJ. A systematic analysis of global anemia burden from 1990 to 2010. Blood. 2014 Jan 30;123(5):615-24. doi: 10.1182/blood-2013-06-508325. Epub 2013 Dec 2. PMID 24297872
- [Background] Zimmermann MB, Hurrell RF. Nutritional iron deficiency. Lancet. 2007 Aug 11;370(9586):511-20. doi: 10.1016/S0140-6736(07)61235-5. PMID 17693180
- [Background] Baumgartner J, Barth-Jaeggi T. Iron interventions in children from low-income and middle-income populations: benefits and risks. Curr Opin Clin Nutr Metab Care. 2015 May;18(3):289-94. doi: 10.1097/MCO.0000000000000168. PMID 25807351
- [Background] Lonnerdal B. Bioactive Proteins in Human Milk: Health, Nutrition, and Implications for Infant Formulas. J Pediatr. 2016 Jun;173 Suppl:S4-9. doi: 10.1016/j.jpeds.2016.02.070. PMID 27234410
- [Background] Manzoni P. Clinical Benefits of Lactoferrin for Infants and Children. J Pediatr. 2016 Jun;173 Suppl:S43-52. doi: 10.1016/j.jpeds.2016.02.075. PMID 27234411
- [Background] Legrand D. Overview of Lactoferrin as a Natural Immune Modulator. J Pediatr. 2016 Jun;173 Suppl:S10-5. doi: 10.1016/j.jpeds.2016.02.071. PMID 27234406
- [Background] Troesch B, Egli I, Zeder C, Hurrell RF, de Pee S, Zimmermann MB. Optimization of a phytase-containing micronutrient powder with low amounts of highly bioavailable iron for in-home fortification of complementary foods. Am J Clin Nutr. 2009 Feb;89(2):539-44. doi: 10.3945/ajcn.2008.27026. Epub 2008 Dec 23. PMID 19106242
- [Background] De-Regil LM, Suchdev PS, Vist GE, Walleser S, Pena-Rosas JP. Home fortification of foods with multiple micronutrient powders for health and nutrition in children under two years of age. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD008959. doi: 10.1002/14651858.CD008959.pub2. PMID 21901727
- [Background] Rai D, Adelman AS, Zhuang W, Rai GP, Boettcher J, Lonnerdal B. Longitudinal changes in lactoferrin concentrations in human milk: a global systematic review. Crit Rev Food Sci Nutr. 2014;54(12):1539-47. doi: 10.1080/10408398.2011.642422. PMID 24580556
- [Background] Liao Y, Jiang R, Lonnerdal B. Biochemical and molecular impacts of lactoferrin on small intestinal growth and development during early life. Biochem Cell Biol. 2012 Jun;90(3):476-84. doi: 10.1139/o11-075. Epub 2012 Feb 14. PMID 22332905
- [Background] Ochoa TJ, Chea-Woo E, Baiocchi N, Pecho I, Campos M, Prada A, Valdiviezo G, Lluque A, Lai D, Cleary TG. Randomized double-blind controlled trial of bovine lactoferrin for prevention of diarrhea in children. J Pediatr. 2013 Feb;162(2):349-56. doi: 10.1016/j.jpeds.2012.07.043. Epub 2012 Aug 30. PMID 22939927
- [Background] Chen K, Chai L, Li H, Zhang Y, Xie HM, Shang J, Tian W, Yang P, Jiang AC. Effect of bovine lactoferrin from iron-fortified formulas on diarrhea and respiratory tract infections of weaned infants in a randomized controlled trial. Nutrition. 2016 Feb;32(2):222-7. doi: 10.1016/j.nut.2015.08.010. Epub 2015 Sep 3. PMID 26602290
- [Background] Chen EZ, Li H. A two-part mixed-effects model for analyzing longitudinal microbiome compositional data. Bioinformatics. 2016 Sep 1;32(17):2611-7. doi: 10.1093/bioinformatics/btw308. Epub 2016 May 14. PMID 27187200

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group A: MMP + Iron + GOS: This study group received daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]) and galacto-oligosaccharides (GOS), 7.5 mg.
  Multiple micronutrient powders with 5 mg iron: The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].
- Study Group B: MMP + Iron + bLF: This study group received daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]), bovine lactoferrin (bLF), 1.0 g.
  Multiple micronutrient powders with 5 mg iron: The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].
- Study Group C: MMP + Iron + GOS + bLF: This study group received daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]), galacto-oligosaccharides (GOS), 7.5 mg, and bovine lactoferrin (bLF), 1.0 g.
  Multiple micronutrient powders with 5 mg iron: The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].
- Study Group D: MMP + Iron: This study group received daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]) alone, with no galacto-oligosaccharides (GOS), and no bovine lactoferrin (bLF).
  Multiple micronutrient powders with 5 mg iron: The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].
Period: Baseline
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Started | 72 | 72 | 72 | 72
Completed | 72 | 72 | 72 | 72
Not Completed | 0 | 0 | 0 | 0
Period: 1 Month Intervention
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Started | 70 | 72 | 70 | 70
Completed | 70 | 72 | 70 | 70
Not Completed | 0 | 0 | 0 | 0
Period: 6 Months Intervention
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Started | 65 | 66 | 65 | 68
Completed | 65 | 66 | 65 | 68
Not Completed | 0 | 0 | 0 | 0
Period: 9 Months Intervention
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Started | 64 | 66 | 65 | 65
Completed | 64 | 66 | 65 | 65
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron | Total
Number analyzed (Participants) | 72 | 72 | 72 | 72 | 288
Age, Continuous [Median (Standard Deviation); unit: months] | 6.07 (0.42) | 6.17 (0.32) | 6.15 (0.37) | 6.27 (0.35) | 6.11 (0.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 36 | 36 | 144
  Male | 36 | 36 | 36 | 36 | 144
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 72 | 72 | 72 | 72 | 288
log(10) Beneficial to Harmful Bacteria Ratio [Mean (Standard Deviation); unit: log(10) ratio] | 2.279 (19.338) | 2.553 (21.663) | 2.070 (17.565) | 1.956 (16.597) | 2.215 (37.582)

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Harmful to Beneficial Bacterial Genera in Fecal Microbiota as Determined by Quantitative Polymerase Chain Reaction (qPCR) at 1 Month
Description: The primary outcome measure will be the ratio of the abundances of potentially harmful (enteropathogenic and/or enterotoxigenic E. coli, C. difficile, members of the C. perfringens group, B. cereus, S. aureus, sum of Shigella spp., and Salmonella) to beneficial (bifidobacteria and the group of Lactobacillus/Leuconostoc/Pediococcus spp.) bacterial genera in fecal microbiota as determined by quantitative polymerase chain reaction (qPCR) at 1 month.
Time Frame: 1 month
Measure: Mean (Standard Error); unit: (unitless)
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 70 | 72 | 70 | 70
(unitless) | 2.208 (0.202) | 1.530 (0.207) | 2.075 (0.220) | 1.292 (0.176)

2. Secondary Outcome: Ratio of Harmful to Beneficial Bacterial Genera in Fecal Microbiota as Determined by Quantitative Polymerase Chain Reaction (qPCR) at 6 Months
Description: A key secondary outcome measure will be the ratio of the abundances of potentially harmful (enteropathogenic and/or enterotoxigenic E. coli, C. difficile, members of the C. perfringens group, B. cereus, S. aureus, sum of Shigella spp., and Salmonella) to beneficial (bifidobacteria and the group of Lactobacillus/Leuconostoc/Pediococcus spp.) bacterial genera in fecal microbiota as determined by quantitative polymerase chain reaction (qPCR) at 6 months.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: (unitless)
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 65 | 66 | 65 | 68
(unitless) | 1.575 (0.169) | 1.699 (0.205) | 1.779 (0.215) | 1.646 (0.200)

3. Secondary Outcome: Ratio of Harmful to Beneficial Bacterial Genera in Fecal Microbiota as Determined by Quantitative Polymerase Chain Reaction (qPCR) at 9 Months
Description: A key secondary outcome measure will be the ratio of the abundances of potentially harmful (enteropathogenic and/or enterotoxigenic E. coli, C. difficile, members of the C. perfringens group, B. cereus, S. aureus, sum of Shigella spp., and Salmonella) to beneficial (bifidobacteria and the group of Lactobacillus/Leuconostoc/Pediococcus spp.) bacterial genera in fecal microbiota as determined by quantitative polymerase chain reaction (qPCR) at 9 months.
Time Frame: 9 months
Measure: Mean (Standard Error); unit: (unitless)
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 64 | 66 | 65 | 65
(unitless) | 2.084 (0.192) | 1.881 (0.183) | 1.916 (0.257) | 1.748 (0.201)

4. Secondary Outcome: Microbiota Composition as Determined by Quantitative Polymerase Chain Reaction (qPCR).
Description: A secondary outcome measure will be the microbiota composition among study groups as determined by quantitative polymerase chain reaction (qPCR) measures of the abundances of potentially harmful (enteropathogenic and/or enterotoxigenic E. coli, C. difficile, members of the C. perfringens group, B. cereus, S. aureus, sum of Shigella spp., and Salmonella) and of beneficial (bifidobacteria and the group of Lactobacillus/Leuconostoc/Pediococcus spp.) bacterial genera at 1, 6, and 9 months. This outcome is reported as the mean log10 fold change from the beneficial to harmful bacteria ratio (BHR) of the baseline microbiota composition, abbreviated as "log10 FC in BHR".
Time Frame: 1, 6 and 9 months
Population: 8 participants in Group A, 6 participants in Group B, 7 participants in Group C, and 7 participants in Group D withdrew during the duration of the study.
Measure: Mean (Standard Error); unit: log 10 (fold change)
Groups:
- Study Group A: MMP + Iron + GOS: This study group will receive daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]) and galacto-oligosaccharides (GOS), 7.5 mg.
  Galacto-oligosaccharides: Galacto-oligosaccharides are classified as Generally Recognized As Safe (GRAS) by the U.S. Food and Drug Administration, are components of cow's milk and have been used repeatedly in clinical trials without adverse effects.
  Multiple micronutrient powders with 5 mg iron: The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].
- Study Group B: MMP + Iron + bLF: This study group will receive daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]), bovine lactoferrin (bLF), 1.0 g.
  Bovine lactoferrin: Bovine lactoferrin is classified as Generally Recognized As Safe (GRAS) by the U.S. Food and Drug Administration, is a component of cow's milk and has been used repeatedly in clinical trials without adverse effects.
  Multiple micronutrient powders with 5 mg iron: The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].
- Study Group C: MMP + Iron + GOS + bLF: This study group will receive daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]), galacto-oligosaccharides (GOS), 7.5 mg, and bovine lactoferrin (bLF), 1.0 g.
  Galacto-oligosaccharides: Galacto-oligosaccharides are classified as Generally Recognized As Safe (GRAS) by the U.S. Food and Drug Administration, are components of cow's milk and have been used repeatedly in clinical trials without adverse effects.
  Bovine lactoferrin: Bovine lactoferrin is classified as Generally Recognized As Safe (GRAS) by the U.S. Food and Drug Administration, is a component of cow's milk and has been used repeatedly in clinical trials without adverse effects.
  Multiple micronutrient powders with 5 mg iron: The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].
- Study Group D: MMP + Iron: This study group will receive daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]) alone, with no galacto-oligosaccharides (GOS), and no bovine lactoferrin (bLF).
  Multiple micronutrient powders with 5 mg iron: The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 72 | 72 | 72 | 72
log 10 (fold change)
  1 month: number analyzed (Participants) | 70 | 72 | 70 | 70
  1 month | -0.022 (0.258) | -1.025 (0.239) | -0.002 (0.314) | -0.637 (0.239)
  6 months: number analyzed (Participants) | 65 | 66 | 65 | 68
  6 months | -0.742 (0.247) | -0.786 (0.291) | -0.308 (0.306) | -0.241 (0.284)
  9 months: number analyzed (Participants) | 64 | 66 | 65 | 65
  9 months | -0.269 (0.290) | -0.607 (0.314) | -0.174 (0.351) | -0.114 (0.284)

5. Secondary Outcome: Number of Participants Who Experienced Diarrhea
Description: A secondary outcome measure will be the prevalence of diarrhea among study groups.
Time Frame: Up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 72 | 72 | 72 | 72
Participants | 7 | 6 | 7 | 4

6. Secondary Outcome: Number of Participants Who Experienced Malaria
Description: A secondary outcome measure will be the prevalence of malaria among study groups.
Time Frame: Up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 72 | 72 | 72 | 72
Participants | 7 | 4 | 3 | 3

7. Secondary Outcome: Proportion of Participants Who Experienced Anemia
Description: A secondary outcome measure will be the proportion of participants with anemia among study groups, defined as Hemoglobin < 11.5 g/L by laboratory diagnosis.
Time Frame: Baseline, 1 month, 6 months, 9 months
Population: as for outcome 4
Measure: Number; unit: Proportion of participants
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 72 | 72 | 72 | 72
Proportion of participants
  Baseline | 0.43 | 0.54 | 0.61 | 0.49
  1 month: number analyzed (Participants) | 70 | 72 | 70 | 70
  1 month | 0.43 | 0.49 | 0.57 | 0.56
  6 months: number analyzed (Participants) | 65 | 66 | 65 | 68
  6 months | 0.35 | 0.33 | 0.31 | 0.31
  9 months: number analyzed (Participants) | 64 | 66 | 65 | 65
  9 months | 0.36 | 0.45 | 0.31 | 0.23

8. Secondary Outcome: Proportion of Participants Who Experienced Iron Deficiency
Description: A secondary outcome measure will be the proportion of participants with iron deficiency among study groups, defined as plasma Ferritin < 12 µg/L or/and soluble transferrin receptor (sTfR) > 8.3 mg/L
Time Frame: Baseline, 1 month, 6 months, 9 months
Population: as for outcome 4
Measure: Number; unit: Proportion of participants
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 72 | 72 | 72 | 72
Proportion of participants
  Baseline | 0.66 | 0.61 | 0.61 | 0.58
  1 month: number analyzed (Participants) | 70 | 72 | 70 | 70
  1 month | 0.3 | 0.3 | 0.39 | 0.37
  6 months: number analyzed (Participants) | 65 | 66 | 65 | 68
  6 months | 0.65 | 0.68 | 0.60 | 0.60
  9 months: number analyzed (Participants) | 64 | 66 | 65 | 65
  9 months | 0.65 | 0.73 | 0.66 | 0.63

9. Secondary Outcome: Proportion of Participants Who Experienced Iron Deficiency Anemia (IDA)
Description: A secondary outcome measure will be the proportion of participants with iron deficiency anemia among study groups, defined as Hemoglobin < 11.5 g/L and Soluble transferrin receptor (sTfR) > 8.3 mg/L
Time Frame: Baseline, 1 month, 6 months, 9 months
Population: as for outcome 4
Measure: Number; unit: Proportion of participants
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 72 | 72 | 72 | 72
Proportion of participants
  Baseline | 0.34 | 0.39 | 0.45 | 0.39
  1 month: number analyzed (Participants) | 70 | 72 | 70 | 70
  1 month | 0.59 | 0.58 | 0.6 | 0.59
  6 months: number analyzed (Participants) | 65 | 66 | 65 | 68
  6 months | 0.29 | 0.30 | 0.22 | 0.26
  9 months: number analyzed (Participants) | 64 | 66 | 65 | 65
  9 months | 0.29 | 0.39 | 0.22 | 0.22

10. Secondary Outcome: Proportion of Participants Who Experienced Inflammation
Description: A secondary outcome measure will be the proportion of participants with inflammation among study groups, defined as C-reactive protein (CRP) > 5 mg/L
Time Frame: Baseline, 1 month, 6 months, 9 months
Population: as for outcome 4
Measure: Number; unit: Proportion of participants
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 72 | 72 | 72 | 72
Proportion of participants
  Baseline | 0.09 | 0.15 | 0.15 | 0.14
  1 month: number analyzed (Participants) | 70 | 72 | 70 | 70
  1 month | 0.12 | 0.11 | 0.13 | 0.14
  6 months: number analyzed (Participants) | 65 | 66 | 65 | 68
  6 months | 0.18 | 0.17 | 0.20 | 0.18
  9 months: number analyzed (Participants) | 64 | 66 | 65 | 65
  9 months | 0.13 | 0.20 | 0.18 | 0.18

11. Secondary Outcome: Number of Participants Who Experienced Respiratory Tract Infections
Description: A secondary outcome measure will be the prevalence of Respiratory tract infections among study groups.
Time Frame: Up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 72 | 72 | 72 | 72
Participants | 40 | 36 | 41 | 38

12. Secondary Outcome: Other Illnesses
Description: A secondary outcome measure will be the prevalence of other illnesses among study groups.
Time Frame: Up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group A: MMP + Iron + GOS | Study Group B: MMP + Iron + bLF | Study Group C: MMP + Iron + GOS + bLF | Study Group D: MMP + Iron
Number analyzed (Participants) | 72 | 72 | 72 | 72
Participants
  Cold | 16 | 10 | 17 | 28
  Dermatitis | 3 | 5 | 2 | 2
  Folliculitis | 2 | 1 | 3 | 4
  Gastritis | 3 | 0 | 7 | 8
  Gastroenteritis | 1 | 3 | 5 | 5
  Impetigo | 3 | 4 | 2 | 5
  Pneumonia | 12 | 3 | 6 | 8
  Rhinitis | 7 | 4 | 3 | 5
  Scabies | 4 | 6 | 6 | 3
  Skin infection | 2 | 5 | 2 | 3
  Tinea capitis | 4 | 3 | 1 | 1

ADVERSE EVENTS:
Time Frame: 9 months
Description: All adverse events reported here represent the clinical (observational) impression of the caregivers.
Groups:
- Study Group D: Iron: This study group will receive daily in-home fortification for 6 months with multiple micronutrient powders with 5 mg iron (as sodium iron EDTA [2.5 mg] and ferrous fumarate [2.5 mg]) alone, with no galacto-oligosaccharides (GOS), and no bovine lactoferrin (bLF).
  Multiple micronutrient powders with 5 mg iron: The multiple micronutrient powders are composed of Vitamin A, 400 μg; Vitamin D, 5 μg; Tocopherol Equivalents, 5 mg; Thiamine, 0.5 mg; Riboflavin, 0.5 mg; Vitamin B6, 0.5 mg; Folic Acid, 90 μg; Niacin, 6 mg; Vitamin B12, 0.9 μg; Vitamin C, 30 mg; Copper, 0.56 mg; Iodine, 90 μg; Selenium, 17 μg; Zinc, 4.1 mg; Phytase, 190 FTU; Iron, 5 mg [(as Ferrous fumarate, 2.5 mg and sodium iron ethylenediaminetetraacetate (NaFeEDTA), 2.5 mg].
Arm/Group | Study Group A: GOS | Study Group B: bLF | Study Group C: GOS + bLF | Study Group D: Iron
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72 | 0/72 | 1/72
Serious Adverse Events (participants affected / at risk) | 1/72 | 1/72 | 0/72 | 1/72
Other Adverse Events (participants affected / at risk) | 56/72 | 55/72 | 59/72 | 65/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group A: GOS (N=72) | Study Group B: bLF (N=72) | Study Group C: GOS + bLF (N=72) | Study Group D: Iron (N=72)
Severe malaria (Infections and infestations) | 1 | 1 | 0 | 0
Hospitalization due to pneumonia (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group A: GOS (N=72) | Study Group B: bLF (N=72) | Study Group C: GOS + bLF (N=72) | Study Group D: Iron (N=72)
Cold (Infections and infestations) | 16 | 10 | 17 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 3 | 4
Cutaneous larva migrans (Infections and infestations) | 0 | 4 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 5 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 7 | 6 | 7 | 4
Fever (General disorders) | 8 | 4 | 4 | 2
Folliculitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 4
Gastritis (Gastrointestinal disorders) | 3 | 0 | 7 | 8
Gastroenteritis (Gastrointestinal disorders) | 1 | 3 | 5 | 5
Impetigo (Infections and infestations) | 3 | 4 | 2 | 5
Malaria (Infections and infestations) | 7 | 4 | 3 | 3
Pneumonia (General disorders) | 12 | 3 | 6 | 8
Rhinitis (General disorders) | 7 | 4 | 3 | 5
Scabies (Skin and subcutaneous tissue disorders) | 4 | 6 | 6 | 3
Skin infection (Infections and infestations) | 2 | 5 | 2 | 3
Tinea capitis (Infections and infestations) | 4 | 3 | 1 | 1
upper respiratory tract infection (URTI) (Respiratory, thoracic and mediastinal disorders) | 40 | 36 | 41 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT03866837/Prot_SAP_000.pdf